CLINICAL TRIAL: NCT02809820
Title: Effects of Selective and Nonselective Beta-blockade on Platelet Aggregation in Patients With Acute Coronary Syndrome
Brief Title: Effects of Beta-blockade on Platelet Aggregation in Acute Coronary Syndrome
Acronym: PLATE-BLOCK
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Giovanni Esposito, MD, PhD, Federico II University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CE-9/14
Record Dates: First submitted 2016-06-20; First posted 2016-06-22 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Acute Coronary Syndrome
Keywords: ACS; Beta Blockers; platelet aggregation; light transmission aggregometry; Beta-Adrenergic Blockers
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Carvedilol; Metoprolol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carvedilol (Active Comparator): Patients who have documented ACS, who are on dual antiplatelet therapy and are randomized to assume carvedilol.
  Interventions: Drug: Carvedilol
- Metoprolol (Active Comparator): Patients who have documented ACS, who are on dual antiplatelet therapy and are randomized to assume metoprolol.
  Interventions: Drug: Metoprolol

INTERVENTIONS:
Drug: Carvedilol — Patients randomized to this group will receive carvedilol at the highest dose tolerated
  Other Names: Selective beta-blocker
  Arms: Carvedilol
Drug: Metoprolol — Patients randomized to this group will receive metoprolol at the highest dose tolerated
  Other Names: Non Selective beta-blocker
  Arms: Metoprolol

SUMMARY:
The Investigators will test the hypothesis that nonselective beta-blockers would have a more pronounced effect on platelet aggregation than selective beta-blockers in patients with acute coronary syndrome treated with dual anti platelet therapy.

DETAILED DESCRIPTION:
In patients with acute coronary syndrome (ACS) beta-blockers are recommended for secondary prevention. It is known that catecholamine levels can potentiate platelet reactivity and beta-blocking agents may also affect platelet aggregation. This effect is mainly mediated by adrenergic receptors on platelets. This suggests that nonselective beta-blockers would have a more pronounced effect on platelet aggregation than selective beta-blockers. However, little is known about the effect of beta-blockers on platelet aggregation in patients with cardiovascular disease and, to date, nothing is known in the setting of ACS.

The aim of the present study is to evaluate the effect of selective and nonselective beta-blockers on platelet aggregation in ACS patients treated with dual anti platelet therapy.

ELIGIBILITY:
Inclusion Criteria:

* Acute Coronary Syndrome
* Current dual anti platelet treatment with acetylsalicylic acid and Ticagrelor

Exclusion Criteria:

* ongoing prasugrel, ticlopidine or clopidogrel therapy
* Creatinine Clearance < 30 ml/min/1.73mm2
* Moderate to severe anemia Hemoglobin < 10 mg/dl
* Platelet count >600000/mm3 or <150000/mm3 or hematocrit >50% or <25%
* concomitant neoplastic or immune-mediated pathologies
* severe pulmonary pathologies
* contraindication to beta blocker therapy.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Platelet aggregation | 30 days
  Platelet aggregation induced by epinephrine is measured by Light Transmission Aggregometry (LTA)

SECONDARY OUTCOMES:
30-days platelet aggregation | 30 days
  Platelet aggregation induced by Adenosine Diphosphate (ADP) is measured by Light Transmission Aggregometry (LTA)
30-days clinical events | 30 days
  Major adverse cardiac events (MACE) and bleedings will be evaluated

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Esposito, MD PhD, Principal Investigator — Federico II University
Locations (1):
- Federico II University of Naples, Naples, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bonten TN, Plaizier CE, Snoep JJ, Stijnen T, Dekkers OM, van der Bom JG. Effect of beta-blockers on platelet aggregation: a systematic review and meta-analysis. Br J Clin Pharmacol. 2014 Nov;78(5):940-9. doi: 10.1111/bcp.12404. PMID 24730697
- [Background] Ignjatovic V, Pavlovic S, Miloradovic V, Andjelkovic N, Davidovic G, Djurdjevic P, Stolic R, Iric-Cupic V, Simic I, Ignjatovic VD, Petrovic N, Smiljanic Z, Zdravkovic V, Simovic S, Jovanovic D, Nesic J. Influence of Different beta-Blockers on Platelet Aggregation in Patients With Coronary Artery Disease on Dual Antiplatelet Therapy. J Cardiovasc Pharmacol Ther. 2016 Jan;21(1):44-52. doi: 10.1177/1074248415581175. Epub 2015 Apr 13. PMID 25868659